CLINICAL TRIAL: NCT03567135
Title: A Retrospective Clinical Study of Postoperative Concurrent Chemoradiotherapy Combined With Anti-angiogenic Drugs in the Treatment of Glioblastoma.
Brief Title: Temozolomide Plus Anti-angiogenesis Drugs and Radiotherapy as a Treatment for Glioblastoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20180524
Record Dates: First submitted 2018-05-30; First posted 2018-06-25 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Glioblastoma
Keywords: Temozolomide; Apatinib; Radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — apatinib; Temozolomide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental 1: concurrent chemoradiotherapy（Temozolomide+apatinib） maintenance therapy（Temozolomide）
  Interventions: Drug: Apatinib; Drug: Temozolomide（TMZ）
- control: concurrent chemoradiotherapy（Temozolomide） maintenance therapy（Temozolomide）
  Interventions: Drug: Temozolomide（TMZ）
- Experimental 2: concurrent chemoradiotherapy（Temozolomide+apatinib） maintenance therapy（Temozolomide+apatinib）
  Interventions: Drug: Apatinib; Drug: Temozolomide（TMZ）

INTERVENTIONS:
Drug: Apatinib — These drugs are planned to inhibit the proliferation and metastasis of tumors.
  Other Names: Temozolomide（TMZ）
  Groups: Experimental 1; Experimental 2
Drug: Temozolomide（TMZ） — Radiotherapy is a common treatment for glioblastoma.Accompanied with TMZ, the damages caused by tumors to the normal tissues will be reduced.

SUMMARY:
Temozolomide (TMZ) is an oral chemotherapy drug. It is an alkylating agent used as a first-line treatment for glioblastoma. This methylation damages the DNA and triggers the death of tumor cells. According to the results of several clinical studies, TMZ synchronous plus radiotherapy and subsequent as adjuvant therapy can significantly improve the survival rate of newly diagnosed glioblastoma patients.

DETAILED DESCRIPTION:
Glioma is the highest incidence of the central nervous system tumor. Surgical treatment is one of the most important therapeutic methods in patients with glioblastoma. But since malignant glioma is a highly invasive tumor, the rate of surgery failure is . So the postoperative therapy shall be accompanied by radiotherapy. Since 1998, the clinical application of Temozolomide(TMZ) has brought hope for malignant glioma patients with its definite curative effect. According to the results of several clinical studies, TMZ synchronous plus radiotherapy and subsequent as adjuvant therapy can significantly improve the survival rate of newly diagnosed GBM patients and break the survival limit of malignant glioma patients. Besides, antiangiogenic therapy is also a choice for the treatment of glioblastoma patients. Vascular endothelial growth factor receptors (VEGFRs) inhibitors block the new formation around the tumor and cut down the supply of oxygen, nutrients and metabolic waste, so that the tumor is hard to proliferate and metastases.

ELIGIBILITY:
Search Criteria:

1. Subjects received anti-angiogenesis drugs simultaneous accompanied with radio-and chemotherapy in Fuzhou Zongyuan since October, 2017;
2. Age: 18-70 years;
3. The first surgical pathology was diagnosed as glioblastoma, WHO grade III or IV;
4. Patients who have previously received no more than one surgical treatment;
5. ECOG performance status: 0-2;
6. Survival expectation≥3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are all previously received anti-angiogenesis drugs simultaneous accompanied with radio-and chemotherapy in Fuzhou Zongyuan since October, 2017.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  in this Survival Duration neither Progression nor death occurs in the subjects.
Assessment of brain edema | From date of randomization until the date of end of the trial, assessed up to 36 months
  The average score of edema grading in patients before and after treatment was calculated separately.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From date of randomization until the date of end of the trial, assessed up to 36 months
  To observe any adverse events that occurred during the clinical study.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided